CLINICAL TRIAL: NCT04753710
Title: A Phase II/III, Randomized, Double-Masked, Vehicle-Controlled, Efficacy, Safety and Tolerability Study of Chloroprocaine 3% Gel Eye Drops in Healthy Volunteers
Brief Title: Efficacy, Safety and Tolerability Study of Chloroprocaine 3% Gel Eye Drops in Healthy Volunteers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sintetica SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHL.3-02-2019
Record Dates: First submitted 2021-01-19; First posted 2021-02-15 (Actual); Results first posted 2022-01-24 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2021-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chloroprocaine (Experimental): Chloroprocaine 3% ocular gel
  Interventions: Drug: Ocular gel
- Placebo (Placebo Comparator): Vehicle for chloroprocaine 3% ocular gel
  Interventions: Drug: Ocular gel

INTERVENTIONS:
Drug: Ocular gel — Instillation

SUMMARY:
The study assess efficacy, safety and tolerability of Chloroprocaine 3% ophthalmic gel in healthy volunteers.

DETAILED DESCRIPTION:
The study is carried out in 2 parts. In part I, safety and tolerability is assessed in three groups (12 subjects per group) for single and multiple instillations (1 drop, 3 drops and 3+3 drops). In each group, 9 subjects is randomized to receive Chloroprocaine 3% Gel and 3 subjects receive vehicle as control in the right eye. After part I is completed, an internal independent board review safety endpoints of data collected from these first subjects and advise to go on with further enrollment.

If no safety concerns arise, in part II efficacy, safety and tolerability is assessed in 60 healthy subjects for the 3 drops dose regimen. 40 subjects receive Chloroprocaine 3% Gel and 20 receive vehicle (2:1 randomization) in the right eye.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent
2. Healthy male or female aged from 18 to 90 years
3. No clinically significant ocular or systemic disease
4. Ability to orally respond to pain
5. Ability to follow the visit schedule

Exclusion Criteria:

Ophthalmic exclusion criteria

1. Eye movement disorder (i.e. Nystagmus)
2. Dacryocystitis and all other pathologies of tears drainage system
3. History of Inflammatory ocular disease (Iritis, uveitis, herpetic keratitis)
4. Corneal, epithelial, stromal or endothelial, residual or evolutionary disease (including corneal ulceration and superficial punctuate keratitis)
5. History of ocular traumatism, infection or inflammation within the last 3 months
6. Best corrected visual acuity < 1/10
7. History of ophthalmic surgical complication (i.e. cystoid macular oedema)

   Systemic/non ophthalmic exclusion criteria
8. General history:

   8.1 Deafness 8.2 Excessive anxiety
9. Any other medical or surgical history, disorder or disease such as acute or chronic severe organic disease: hepatic, endocrine neoplastic, haematological diseases, severe psychiatric illness, relevant cardiovascular abnormalities (such as unstable angina, uncontrolled hypertension: systolic blood pressure over 200 mm Hg, diastolic blood pressure over 100 mm Hg) and/or any complicating factor or structural abnormality judged by the investigator to be incompatible with the study
10. Allergic history: Known hypersensitivity to one of the components of the study medications or to test products

    Specific non-inclusion criteria for women:
11. Pregnancy, lactation
12. Women without an effective method of contraception (i.e. oral contraceptive, intra-uterine device, subcutaneous contraceptive implant) OR
13. Women not hysterectomised, not menopausal nor surgically sterilized

    Exclusion criteria related to general conditions:
14. Inability of subject to understand the study procedures and thus inability to give informed consent
15. Non-compliant subject (e.g. not willing to attend the follow-up visits, way of life interfering with compliance)
16. Participation in another clinical study
17. Already included once in this study
18. Ward of court
19. Subject not covered by the Social Security

    Exclusion criteria related to previous and concomitant medications (taken within 15 days prior screening visit)
20. Use of systemic opioids and opioid drugs
21. Topical ocular treatment with anaesthetic action
22. Use of systemic analgesic drugs (except paracetamol, which will be allowed after Visit 2)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhoefer, Principal Investigator — Universitätsklinik für Klinische Pharmakologie
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In part 1: 36 subjects received treatment and completed the study. in part 2: 60 were randomized, 40 in the CHL 3% gel and 20 in the vehicle group.
Period: Overall
Arm/Group | Chloroprocaine | Placebo
Started | 67 | 29
Completed | 67 | 29
Not Completed | 0 | 0
Period: First Phase
Arm/Group | Chloroprocaine | Placebo
Started | 27 | 9
Completed | 27 | 9
Not Completed | 0 | 0
Period: Second Phase
Arm/Group | Chloroprocaine | Placebo
Started | 40 | 20
Completed | 40 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chloroprocaine | Placebo | Total
Number analyzed (Participants) | 67 | 29 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (5.4) | 25.7 (5.5) | 25.6 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 16 | 52
  Male | 31 | 13 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 67 | 29 | 96

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Phase 2 With Anesthesia Success
Description: Estimate the proportion of subjects experiencing full anaesthesia of the ocular surface 5 minutes after administration of Chloroprocaine 3% ophthalmic gel (the intent was to collect and only report data for Participants who were in Phase 2)
Time Frame: Day 1
Measure: Number; unit: participants
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 40 | 20
participants
  Anesthesia success | 38 | 4
  No success | 2 | 16

2. Secondary Outcome: Duration of Anesthesia Only in Patients in Phase 2
Description: Duration of anesthesia (min) for subjects in phase 2 (the intent was to collect and only report data for Participants who were in Phase 2)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 40 | 20
minutes | 24.15 (8.83) | 19.3 (14.72)

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Ocular symptoms and Adverse events
Time Frame: Up to 29 days
Measure: Number; unit: participants
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 67 | 29
participants | 43 | 15

4. Secondary Outcome: Mean Arterial Pressure
Description: Mean arterial pressure (mmHg) is defined as the average pressure in a patient's arteries during one cardiac cycle. It is considered a better indicator of perfusion to vital organs than systolic blood pressure (SBP).
Time Frame: up to 8 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 67 | 29
mmHg
  Visit 1 Screening | 95 (9) | 94 (9)
  Visit 2 pre-dose | 96 (8) | 94 (9)
  Visit 2 post-dose | 95 (8) | 92 (9)
  Visit 4 Follow-up | 95 (8) | 94 (9)

5. Secondary Outcome: Number of Participants With Anomalies in Slip Lamp Examination
Description: Number of Participants with Anomalies in Slip Lamp Examination
Time Frame: up to 8 days
Measure: Number; unit: participants
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 67 | 29
participants | 17 | 5

6. Secondary Outcome: Number of Participants With Anomalies in Corneal Fluorescein Staining
Description: Number of Participants with anomalies found with corneal fluorescein staining
Time Frame: up to 8 days
Measure: Number; unit: participants
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 67 | 29
participants | 0 | 0

7. Secondary Outcome: Ocular Pressure
Description: Intraocular pressure (mmHg)
Time Frame: Follow up (up to 8 days)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 67 | 29
mmHg
  screening | 14 (2.6) | 14 (2.3)
  follow up | 13.6 (2.6) | 13.3 (2)

ADVERSE EVENTS:
Time Frame: Study duration (Up to 29 days)
Arm/Group | Chloroprocaine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/29
Other Adverse Events (participants affected / at risk) | 43/67 | 15/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chloroprocaine (N=67) | Placebo (N=29)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
bradycardia (Cardiac disorders) | 5 (5) | 0 (0)
Conjunctival hemorrhage (Eye disorders) | 0 (0) | 2 (2)
Conjunctival edema (Eye disorders) | 1 (1) | 0 (0)
dry eye (Eye disorders) | 1 (1) | 0 (0)
eye irritation (Eye disorders) | 7 (7) | 2 (2)
mydriasis (Eye disorders) | 23 (23) | 1 (1)
ocular hyperemia (Eye disorders) | 1 (1) | 0 (0)
vision blurred (Eye disorders) | 3 (3) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 1 (1) | 0 (0)
instillation site pain (General disorders) | 1 (1) | 0 (0)
pain (General disorders) | 1 (1) | 0 (0)
Sensation of foreign body (General disorders) | 3 (3) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0)
Sars-cov-2 test positive (Investigations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 4 (4)
presyncope (Nervous system disorders) | 0 (0) | 1 (1)
syncope (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT04753710/Prot_SAP_000.pdf